CLINICAL TRIAL: NCT03337555
Title: A Comparison of McGrath MAC®, Pentax-AWS® and Macintosh Direct Laryngoscopes for Nasotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Clinical assitant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AJIRB-MED-OBS-17-327
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Intubation;Difficult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Macintosh (Active Comparator): intubation using Macintosh direct laryngoscope
  Interventions: Device: Macintosh
- McGrath (Experimental): intubation using McGrath MAC®
  Interventions: Device: McGrath
- Pentax (Experimental): intubation using Pentax-airway scope®
  Interventions: Device: Pentax

INTERVENTIONS:
Device: McGrath — McGrath videolaryngoscope
  Arms: McGrath
Device: Pentax — Pentax videolaryngoscope
  Arms: Pentax
Device: Macintosh — Macintosh direct laryngoscope
  Arms: Macintosh

SUMMARY:
A comparison of intubation time, difficulty of intubation in nasotracheal intubation using McGrath MAC®, Pentax-AWS® and Macintosh direct laryngoscopes

DETAILED DESCRIPTION:
This trial is prospective randomized trial. The Objects are adult patients who need nasotracheal intubation for surgery. Using computed randomized table, participants are assigned to three groups, McGrath MAC®, Pentax-AWS® and Macintosh direct laryngoscopes.

The intubation will be done by One expert anesthesiologist who have more than 10 years experience.

Investigators compare intubation time, success rate and difficulty between three groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 19 years old
* ASA I or II
* Patients who need nasotracheal intubation for surgery

Exclusion Criteria:

* Anatomical deformity in head and neck
* Modified Mallampati score IV
* Bleeding tendency in preoperative evaluation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Intubation time | within 5 minutes
  from endotracheal tube pass the nostril to end-tidal CO2 appear

SECONDARY OUTCOMES:
Success rate | within 5 minutes
  Failure defined intubation time more than 120sec or SaO2 less than 95%

CONTACTS AND LOCATIONS:
Overall Officials: Yun Jeong Chae, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university schoole of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No